CLINICAL TRIAL: NCT04352777
Title: Evaluation of the Effects of Endocrine Therapy and Abemaciclib on Host and Tumor Immune Cell Repertoire/Function in Advanced ER+/HER2- Breast Cancer
Brief Title: Impact of Endocrine Therapy and Abemaciclib on Host and Tumor Immune Cell Repertoire/Function in Advanced ER+/HER2- Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103625
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Breast Cancer; Locally Advanced Breast Cancer; Hormone Receptor Positive Tumor
Keywords: metastatic breast cancer; abemaciclib; endocrine therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Fulvestrant; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Active Comparator): Fulvestrant plus abemaciclib
  Interventions: Drug: Abemaciclib; Drug: Fulvestrant
- Cohort 2 (Active Comparator): Aromatase inhibitor plus abemaciclib (with or without ovarian suppression)
  Interventions: Drug: Abemaciclib; Drug: Aromatase Inhibitors

INTERVENTIONS:
Drug: Abemaciclib — 50 - 150mg tablet BID as prescribed per standard of care
Drug: Fulvestrant — 500mg as prescribed per standard of care
  Arms: Cohort 1
Drug: Aromatase Inhibitors — Letrozole, anastrozole as prescribed per standard of care
  Arms: Cohort 2

SUMMARY:
The purpose of this study is to perform an in depth analysis of changes in the tumor immune microenvironment in patients undergoing treatment with standard of care endocrine therapy and abemaciclib in the advanced setting via singe cell RNA sequencing. The investigators will also correlate changes in serum estrogen levels to changes in tumor and peripheral immune cell repertoire and function (including regulatory T cell populations, B cells, myeloid-derived suppressor cell populations, T cell activation and T cell exhaustion).This study has two cohorts with 15 patients in each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Women age ≥ 18
2. Locally advanced/unresectable or metastatic breast cancer
3. Histologically documented estrogen receptor positive adenocarcinoma of the breast that is (any progesterone status allowed):

   * ER positive defined as ≥ 10 % tumor cells positive for ER by immunohistochemistry (IHC), irrespective of staining intensity.
   * HER2 negative status is determined by:
   * IHC 1+, as defined by incomplete membrane staining that is faint/barely perceptible and within > 10% of invasive tumor cells, or
   * IHC 0, as defined by no staining observed or membrane staining that is incomplete and is faint/barely perceptible and within ≤ 10% of the invasive tumor cells, or
   * FISH negative based on:
   * Single-probe average HER2 copy number < 4.0 signals / cell, or
   * Dual-probe HER2/CEP17 ratio < 2.0 with an average HER2 copy number < 4.0 signals /cell
4. Patients should have plans to initiate standard of care endocrine therapy with non-steroidal aromatase inhibitor (letrozole, anastrazole) OR fulvestrant plus abemaciclib in the advanced/metastatic first-line or second-line setting per treating oncologist discretion
5. Patients should be willing and able to undergo fresh biopsy pretreatment and at 4 weeks into treatment.
6. Patients should have an accessible lesion representative of recurrent or metastatic breast cancer for biopsy. Patients will undergo a tissue biopsy or tissue collection for research purposes only. Sites for tissue acquisition include the breast, skin/chest wall, soft tissue, liver, bone. Research directed lung biopsies and brain biopsies are not permitted. Procedures for tissue acquisition are restricted to those performed under local anesthesia or IV conscious sedation; biopsies that require general anesthesia are not permitted in this situation.
7. Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to randomization. A washout period of at least 21 days is required between last chemotherapy dose and randomization (provided the patient did not receive radiotherapy).
8. Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy.
9. The patient is able to swallow oral medications.
10. The patient has adequate organ function for all of the following criteria, as defined in below.

    * Hematologic
    * ANC ≥1.5 × 10^9/L
    * Platelets ≥100 × 10^9/L
    * Hemoglobin ≥ 8 g/dL. * Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.
    * Hepatic
    * Total bilirubin ≤1.5 × ULN *Patients with Gilbert's syndrome with a total bilirubin ≤ 2.0 times ULN and direct bilirubin within normal limits are permitted.
    * ALT and AST ≤ 3 × ULN

      * Abbreviations: ALT = alanine aminotransferase; ANC = absolute neutrophil count; AST = aspartate aminotransferase; ULN = upper limit of normal.
11. Able and willing to complete the informed consent process
12. Agree to have bio-specimens stored for future research

Exclusion Criteria:

1. History of concurrent active malignancy within last 5 years (excluding basal cell skin cancer, resected squamous cell carcinoma of the skin)
2. Current use of hormonal birth control (copper IUD allowed) or estrogen replacement therapy
3. Active autoimmune disease that has required systemic treatment in past 6 months (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or similar treatment) is not considered a form of systemic treatment.
4. History of a serious or life-threatening allergic reaction to local anesthetics (e.g., lidocaine, xylocaine) used during a biopsy procedure
5. Immunodeficient subjects, E.G., receiving systemic steroid therapy greater than physiologic doses or any other form of immunosuppressive therapy within 30 days prior to the first dose of endocrine therapy treatment
6. Concurrent use of other oncologic therapies in the adjuvant setting other than bisphosphonates
7. Patients with disease not amenable to biopsy
8. The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
9. Females who are pregnant or lactating.
10. The patient has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
11. The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
12. History of bleeding disorder that would make serial biopsies unsafe.
13. Patients of active anticoagulation for history of venous thromboembolism, cardiovascular conditions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Changes in serum estrogen (E1 and E2) levels compared to changes in tumor immune cell repertoire and function in response to endocrine therapy and CDK 4/6 inhibition | Through study completion, approximately 2 years
  Estrogen levels in the blood will be assessed to correlate with changes in immune cell populations within the tumor.
Changes in serum estrogen (E1 and E2) levels compared to peripheral blood mononuclear cell repertoire and function in response to endocrine therapy and CDK 4/6 inhibition | Through study completion, approximately 2 years
  Estrogen levels in the blood will be assessed to correlate with changes in the characterization and functionality of peripheral blood mononuclear cells including regulatory T cell populations, B cells, myeloid-derived suppressor cell populations, T cell activation and T cell exhaustion.

SECONDARY OUTCOMES:
Changes in tumor immune cell populations in response to fulvestrant and aromatase inhibitor therapy plus abemaciclib, measured by sequential biopsies | Baseline, 4 weeks
  Changes in tumor immune cell populations will be assessed by sequential biopsies via single cell RNA sequencing analysis of fresh tissue
Differences in tumor immune cell infiltrate and peripheral blood mononuclear cells in response to fulvestrant versus aromatase inhibition plus CDK4/6 inhibition, measured by sequential biopsies and blood collection | Baseline, 4 weeks
  Tumor immune cell and peripheral blood monoclonal cell changes assessed by sequential biopsies via single cell RNA sequencing analysis of fresh tissue
To correlate unique immune cell populations identified with progression free survival in the overall population | Through study completion, approximately 2 years
  Unique immune cell populations will be identified via single cell RNA sequencing and correlated to progression free survival measured by RECIST1.1.
Best overall response rate of abemaciclib and endocrine therapy in both treatment arms | Through study completion, approximately 2 years
  Best overall response rate to both treatment arms measured by RECIST 1.1
Progression free survival in response to abemaciclib and endocrine therapy in both treatment arms | Through study completion, approximately 2 years
  Progression free survival rate to both treatment arms measured by RECIST 1.1
Number of participants with at least one serious adverse event | Through study completion, approximately 2 years
  Serious adverse events will include only those related to abemaciclib, endocrine therapy, and/or study-related biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Sammons, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No